CLINICAL TRIAL: NCT06855264
Title: A Phase 1, Randomized, Single-Dose, Positive- and Placebo-Controlled, 3-Way Crossover Study to Evaluate the Effects of Varegacestat on Cardiac Repolarization in Healthy Participants
Brief Title: A Cardiac Liability Study of Varegacestat in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immunome, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: AL102-502
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
Keywords: thorough-QT
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) This is a double-blind study (with respect to varegacestat and placebo only; moxifloxacin will be open label).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Varegacestat (Experimental)
  Interventions: Drug: varegacestat
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: varegacestat — Single oral dose of varegacestat
  Arms: Varegacestat
Drug: Placebo — Single oral dose of placebo
  Arms: Placebo
Drug: Moxifloxacin 400 mg — Single oral dose of moxifloxacin
  Arms: Moxifloxacin

SUMMARY:
This clinical study is designed to study the effect of a single dose of varegacestat on cardiac repolarization in healthy adult participants.

DETAILED DESCRIPTION:
This is a double-blind (with respect to varegacestat and placebo only), single-dose, randomized, placebo- and positive- controlled, 3-way crossover study.

On Day 1 of each period, participants will receive one of 3 treatments: a single dose of varegacestat (Treatment A), a single dose of varegacestat matching placebo (Treatment B), or a single dose of moxifloxacin (Treatment C). In each period, cardiodynamic ECGs will be collected predose and for 24 hours postdose. PK samples will be collected predose and up to 168 hours post-dose for assessments of varegacestat and AL102 MTB, and up to 24 hours post-dose for assessment of moxifloxacin.

There will be a washout of at least 14 days between doses. Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female (of non childbearing potential), 18 to 55 years of age, inclusive, at the screening visit.
* Medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, and vital signs, as deemed by the PI or designee

Exclusion Criteria:

* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or pose an additional risk to the participant by their participation in the study.
* Have taken an investigational drug or participated in a clinical trial evaluating an investigational drug or device within 30 days (or 5 half-lives) prior to the study drug dose, whichever is longer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected change from baseline QTc and varegacestat and its metabolite, AL102 MTB, plasma concentrations | 24 hours

SECONDARY OUTCOMES:
Change from baseline, placebo-corrected, and categorical outliers of the ECG parameter HR from a single oral dose of varegacestat. | 24 hours
Change from baseline and placebo-corrected ECG parameter QT from a single oral dose of varegacestat. | 24 hours
Change from baseline, placebo-corrected, and categorical outliers of the ECG parameter QTcF from a single oral dose of varegacestat. | 24 hours
The AUC from time 0 extrapolated to infinity, calculated as the sum of AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant of varegacesatat and AL102-MTB (varegacestat metabolite). | 7 days
Maximum observed concentration (Cmax) of varegacesatat and AL102-MTB (varegacestat metabolite). | 7 days
Apparent first-order terminal elimination half-life (t1/2) will be calculated as 0.693/Kel of varegacesatat and AL102-MTB (varegacestat metabolite). | 7 days
Safety and tolerability of a single oral dose of varegacestat by incidences of treatment-emergent adverse events. | Approximately 56 days
Assay sensitivity of the study to detect a small QTc effect using moxifloxacin as a positive control. | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided